CLINICAL TRIAL: NCT06462105
Title: Randomized Phase II Clinical Study of Liposomal Irinotecan or Etoposide Combined With Carboplatin and Serplulimab as First-line Treatment for Extensive Stage Small Cell Lung Cancer
Brief Title: Liposomal Irinotecan Combination Regimen for First-line Treatment of Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhou Chengzhi (Other)
Collaborators: Sun Yat-sen University (Other); Hunan Cancer Hospital (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); First People's Hospital of Foshan (Other); Youjiang Medical College for Nationalities (Other)
Responsible Party: Sponsor-Investigator, Zhou Chengzhi, Health technician, Guangzhou Institute of Respiratory Disease
Organization: Guangzhou Institute of Respiratory Disease (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ES-2024-072-02
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liposomal irinotecan + Carboplatin + Serplulimab (Experimental): Liposomal irinotecan: 50mg/m2, ivgtt, d1; Carboplatin AUC=5, ivgtt, d1; Serplulimab: 4.5mg/kg, ivgtt, d1; The drug was administered once every three weeks for a total of 4 cycles. After 4 cycles, serplulimab is maintained until disease progression or toxicity becomes intolerable.
  Interventions: Drug: Irinotecan Hydrochloride Liposome Injection；Carboplatin Injection；Serplulimab Injection
- Etoposide + Carboplatin + Serplulimab (Experimental): Etoposide: 100 mg/m2, ivgtt, d1-3; Carboplatin AUC=5, ivgtt, d1; Serplulimab: 4.5mg/kg, ivgtt, d1; The drug was administered once every three weeks for a total of 4 cycles. After 4 cycles, serplulimab is maintained until disease progression or toxicity becomes intolerable.
  Interventions: Drug: Irinotecan Hydrochloride Liposome Injection；Carboplatin Injection；Serplulimab Injection

INTERVENTIONS:
Drug: Irinotecan Hydrochloride Liposome Injection；Carboplatin Injection；Serplulimab Injection — Cohort 1: Liposomal irinotecan: 50mg/m2, ivgtt, d1; Carboplatin AUC=5, ivgtt, d1; Serplulimab: 4.5mg/kg, ivgtt, d1; The drug was administered once every three weeks for a total of 4 cycles. After 4 cycles, serplulimab is maintained until disease progression or toxicity becomes intolerable.
  Cohort 2: Etoposide: 100 mg/m2, ivgtt, d1-3; Carboplatin AUC=5, ivgtt, d1; Serplulimab: 4.5mg/kg, ivgtt, d1; The drug was administered once every three weeks for a total of 4 cycles. After 4 cycles, serplulimab is maintained until disease progression or toxicity becomes intolerable.
  Other Names: Etoposide Injection；Carboplatin Injection；Serplulimab Injection

SUMMARY:
Lung cancer is a malignant tumor with high incidence and mortality in China and the world, among which small cell lung cancer (SCLC) accounts for 13% to 17% of lung cancer, and about 250,000 patients are diagnosed with SCLC every year in the world, and nearly 200,000 people die from it. Due to the high degree of malignancy of SCLC, it is easy to develop distant metastasis in the early stage, and most of the patients are diagnosed in the late stage with poor prognosis. Although SCLC is sensitive to chemotherapy and radiotherapy and has a high remission rate after initial treatment, it is prone to secondary drug resistance and relapse. SCLC is a low-differentiated, high-grade neuroendocrine tumor that can be classified into limited-stage and extensive stage (ES-SCLC). Etoposide combined with cisplatin (EP regimen) or carboplatin (EC regimen), irinotecan combined with cisplatin (IP regimen) or carboplatin (IC regimen) are the basis of standard first-line therapy for ES-SCLC. Immunocombined chemotherapy has also become the first-line standard treatment for ES-SCLC, among which serplulimab + etoposide + carboplatin is recommended by CSCO guidelines for first-line treatment. Liposomal irinotecan is irinotecan encapsulated by liposomes, which has advantages in safety. The study is expected to achieve good efficacy, improve the quality of life and prolong the survival of patients by combining the immune drug serplulimab on the basis of IC regimen. After replacing ordinary irinotecan with liposomal irinotecan, this study aims to compare the efficacy and safety of liposomal irinotecan + carboplatin + serplulimab with the first-line standard regimen (etoposide + carboplatin + serplulimab) in patients with extensive stage small-cell lung cancer, providing a better basis for clinical use.

DETAILED DESCRIPTION:
Lung cancer is a malignant tumor with high incidence and mortality in China and the world, among which small cell lung cancer (SCLC) accounts for 13% to 17% of lung cancer, and about 250,000 patients are diagnosed with SCLC every year in the world, and nearly 200,000 people die from it. Due to the high degree of malignancy of SCLC, it is easy to develop distant metastasis in the early stage, and most of the patients are diagnosed in the late stage with poor prognosis. Although SCLC is sensitive to chemotherapy and radiotherapy and has a high remission rate after initial treatment, it is prone to secondary drug resistance and relapse. SCLC is a low-differentiated, high-grade neuroendocrine tumor that can be classified into limited-stage and extensive stage (ES-SCLC). Etoposide combined with cisplatin (EP regimen) or carboplatin (EC regimen), irinotecan combined with cisplatin (IP regimen) or carboplatin (IC regimen) are the basis of standard first-line therapy for ES-SCLC. Immunocombined chemotherapy has also become the first-line standard treatment for ES-SCLC, among which serplulimab + etoposide + carboplatin is recommended by CSCO guidelines for first-line treatment. Liposomal irinotecan is irinotecan encapsulated by liposomes, which has advantages in safety. The study is expected to achieve good efficacy, improve the quality of life and prolong the survival of patients by combining the immune drug serplulimab on the basis of IC regimen. After replacing ordinary irinotecan with liposomal irinotecan, this study aims to compare the efficacy and safety of liposomal irinotecan + carboplatin + serplulimab with the first-line standard regimen (etoposide + carboplatin + serplulimab) in patients with extensive stage small-cell lung cancer, providing a better basis for clinical use.

Trial design: This is a multicenter, open-label, non-comparative, randomized Phase II clinical study. Sixty patients with extensive stage small cell lung cancer were expected to be enrolled and randomly assigned 1:1 to either liposomal irinotecan + carboplatin + serplulimab or etoposide + carboplatin + serplulimab for treatment. The study included a screening period (within 28 days), a treatment period (4 cycles planned), and a follow-up period (safety follow-up and PFS follow-up). Subjects signed informed consent and underwent baseline examination during the screening period. Patients who met the inclusion and exclusion criteria entered the treatment period. All subjects completed relevant examinations specified in the protocol during treatment to observe safety, tolerability and efficacy. The same subject received only one dosing schedule during the study. After the treatment period, the follow-up period was entered.

Treatment regimen: Cohort 1: Liposomal irinotecan: 50mg/m2, ivgtt, d1; Carboplatin AUC=5, ivgtt, d1; Serplulimab: 4.5mg/kg, ivgtt, d1; The drug was administered once every three weeks for a total of 4 cycles. After 4 cycles, serplulimab is maintained until disease progression or toxicity becomes intolerable. Cohort 2: Etoposide: 100 mg/m2, ivgtt, d1-3; Carboplatin AUC=5, ivgtt, d1; Serplulimab: 4.5mg/kg, ivgtt, d1; The drug was administered once every three weeks for a total of 4 cycles. After 4 cycles, serplulimab is maintained until disease progression or toxicity becomes intolerable.

Endpoint: Primary endpoint: Progression-free survival (PFS). Secondary endpoints: Objective response rate (ORR), disease control rate (DCR), overall survival (OS), and outcome in brain metastases (PFS).

Safety endpoints: Incidence and severity of hematologic and nonhematologic adverse events (NCI-CTCAE5.0).

Follow-up: After the end of the treatment period, the follow-up period was entered, which was once every 2 months in the first year and once every 3-4 months in the second to third year.

Statistical analysis: IBM SPSS software (version 25.0 or above) was used for statistical analysis in this study. The measurement data were described statistically with mean, median, standard deviation, maximum and minimum values. Count data or grade data use case number, percentage representation.

ELIGIBILITY:
Inclusion Criteria:

* Patients fully understand the study, voluntarily participate and sign an informed consent form (ICF)；
* Age ≥18 years；
* Patients with pathologically or histologically confirmed extensive stage small cell Lung cancer (according to the Veterans Administration Lung Study Group, VALG staging system)；
* The patient had not previously received any form of antitumor therapy；
* According to RECIST1.1 criteria, the patient had at least one measurable target lesion；
* Eastern Cooperative Oncology Group（ECOG）Physical status score: 0-2；
* The expected survival time is ≥3 months；
* Absolute neutrophil count (ANC) ≥1.5×10^9/L, platelets ≥100×10^9/L, and hemoglobin ≥90 g/L (no blood transfusion, blood products, correction with granulocyte colony stimulating factor or other hematopoietic stimulating factor within 14 days prior to laboratory examination)；
* Serum creatinine ≤1.5 times the upper limit of normal value; AST and ALT ≤2.5 times the upper limit of normal (≤5 times the upper limit of normal for patients with liver invasion); Total bilirubin ≤1.5 times the upper limit of normal (≤3 times the upper limit of normal for patients with liver invasion)；
* Women of childbearing age must have had a pregnancy test (serological) negative within 7 days prior to enrollment and be willing to use an appropriate method of contraception during the trial period and for 6 months after the last dose of the test drug.

Exclusion Criteria:

* Patients with large cell neuroendocrine tumor and mixed small cell carcinoma；
* Patients with active brain metastases or central nervous system invasion； confirmed by imaging evaluation and/or biopsy (prednisone equivalent dose ≥10mg)；
* Allergic reaction to any investigational drug or its ingredients；
* The patient has previously received other antibodies/drugs that target immune checkpoints, such as PD-1, PD-L1, CTLA4, etc；
* Serious, uncontrolled comorbidities that could affect the study results, including but not limited to serious infections, diabetes, or cardiovascular and cerebrovascular disease, were identified；
* Imaging confirmed intestinal obstruction；
* It has uncontrollable ascites, abdominal infection and pyloric obstruction；
* Cardiac function and disease: a history of myocardial infarction, unstable angina pectoris, severe unstable ventricular arrhythmia or any other arrhythmia requiring treatment, a history of clinically serious pericardial disease, or electrocardiographic evidence of acute ischemic or active conduction system abnormalities in the 6 months prior to recruitment；
* Hepatitis B, hepatitis C active infection (hepatitis B surface antigen positive and hepatitis B DNA more than 1x103 copies /mL; more than 1x103 copies /mL of HCV RNA)；
* Human immunodeficiency virus (HIV) infection (HIV antibody positive);
* Previous or current co-occurrence of other malignancies (in addition to non-melanoma basal cell carcinoma of the skin that is effectively controlled, breast/cervical carcinoma in situ, and other malignancies that have been effectively controlled without treatment within the past five years);
* Pregnant and lactating women and patients of childbearing age who do not want to use contraception;
* The investigators determined that patients were not suitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-05 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival（PFS） | The time between the subject's signing of the informed consent and the onset of tumor progression (according to RECIST v1.1 criteria) or death.
  The PFS will be analyzed using Kaplan-Meier method and 95% bilateral confidence intervals will be calculated

SECONDARY OUTCOMES:
Objective response rate（ORR） | Percentage of tumor volume reduction to complete response (CR) and partial response (PR) (according to RECIST v1.1 criteria).
  ORR use cases, percentage representation
Disease control rate（DCR） | Best tumor response based on RECIST1.1 criteria, the proportion of CR, PR and SD.
  DCR use cases, percentage representation
Overall survival（OS） | The time between the subject signing the informed consent form and the patient's death due to various causes.
  The OS will be analyzed using Kaplan-Meier method and 95% bilateral confidence intervals will be calculated
Incidence and severity of hematological and non-hematological adverse events | The time between the subject signing the informed consent and the end of treatment
  Safety: The number and frequency of adverse events, serious adverse events, and treatment-related adverse events (NCI CTCAE v5.0) individually and collectively were listed and the incidence rate was calculated.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code